CLINICAL TRIAL: NCT02819492
Title: Side Specific Withdrawal Times for Colonoscopy: Impact on Adenoma Detection in the Proximal and Distal Colon
Acronym: SNOWCAT
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: SNOWCAT
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2016-10

CONDITIONS: Colon Adenoma
Keywords: Adenoma; Colonoscopy; Withdrawal; Proximal; Observation Time
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Colon polyps
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Routine colonoscopy Cohort: Patients receiving routine colonoscopy at the study site

SUMMARY:
Adenoma detection in the main goal of screening colonoscopy. In order to detect adenomas it is mandatory to spend a long enough time investigating the colonic mucosa. A minimum observation time of 6 minutes has been proposed as a quality criterion for screening colonoscopy. However, different locations of the colon (proximal, distal) may require specific observation time periods. The colon can be divided into a proximal (right) and distal (left) part. Until now, it is unclear whether observation time has a significant impact on adenoma detection in both parts of the colon. The aim of this study therefore is to conduct a trial in which side-specific observation times and adenoma detection rates are measured in order to investigate this correlation in particular for the right colon.

ELIGIBILITY:
Inclusion Criteria:

* indication for colonoscopy
* age ≥ 40 years

Exclusion Criteria:

* American Society of Anesthesiologists class IV or higher
* pregnant women
* indication for colonoscopy: inflammatory bowel disease
* indication for colonoscopy: polyposis syndrome
* indication for colonoscopy: emergency colonoscopy e.g. acute bleeding
* contraindication for polyp resection e.g. patients on warfarin

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving colonoscopy at the study site are eligible for participation.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-11; Primary Completion 2016-10 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate in the proximal colon | up to 2 weeks (participants will be followed for the duration of hospital stay or outpatient treatment, an expected average of 2 weeks)
  After obtaining the histopathological diagnosis of resected polyps (approximately 3 -6 days) it can be determined whether the resected polyp contained adenomatous histology or not.

SECONDARY OUTCOMES:
Polyp detection rate | up to one day
  a maximum of one day is expected for colonoscopy procedures

CONTACTS AND LOCATIONS:
Locations (1):
- II Medizinische Klinik am Klinikum rechts der Isar der Technischen Universität München, Munich, Germany

IPD SHARING:
Plan to Share IPD: No